CLINICAL TRIAL: NCT02847494
Title: Corticosteroids for Acute Migraine. An ED-based, Randomized, Comparative Effectiveness Trial
Brief Title: Corticosteroids for Acute Migraine in the Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, PI, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2016-6342
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Metoclopramide; Dexamethasone; Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Metoclopramide 10mg IV+ dexamethasone 10mg IM
  Interventions: Drug: metoclopramide; Drug: Dexamethasone
- Experimental (Active Comparator): Metoclopramide 10mg IV + methylprednisolone acetate 160mg IM
  Interventions: Drug: metoclopramide; Drug: methylprednisolone acetate

INTERVENTIONS:
Drug: metoclopramide — metoclopramide 10mg intravenous infusion over 15 minutes
Drug: Dexamethasone — dexamethasone 10mg intramuscular injection
  Arms: Control
Drug: methylprednisolone acetate — methylprednislone acetate 160mg intramuscular injection
  Arms: Experimental

SUMMARY:
This is an emergency department based randomized trial in which we compare two different treatment for migraine headache. The goal is to decrease the number of headache days during the week after ED discharge.

ELIGIBILITY:
Inclusion Criteria:

* Migraine without aura criteria (International Classification of Headache Disorders 3B )
* Headache rated as moderate or severe in intensity

Exclusion Criteria:

* Concern for secondary cause of headache
* Contra-indications to investigational medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2017-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Friedman, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - Montefiore Medical Center--Einstein, The Bronx, New York
  - Montefiore Medical Center-Moses, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Latev A, Friedman BW, Irizarry E, Solorzano C, Restivo A, Chertoff A, Zias E, Gallagher EJ. A Randomized Trial of a Long-Acting Depot Corticosteroid Versus Dexamethasone to Prevent Headache Recurrence Among Patients With Acute Migraine Who Are Discharged From an Emergency Department. Ann Emerg Med. 2019 Feb;73(2):141-149. doi: 10.1016/j.annemergmed.2018.09.028. Epub 2018 Nov 16. PMID 30449536

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Experimental
Started | 109 | 111
Completed | 101 | 106
Not Completed | 8 | 5
Not completed — Lost to Follow-up | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 109 | 111 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (13) | 39 (16) | 38 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 94 | 187
  Male | 16 | 17 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 109 | 111 | 220
Duration of headache [Median (Inter-Quartile Range); unit: hours] | 48 [24 to 96] | 72 [24 to 120] | 72 [24 to 96]

OUTCOME MEASURES:

1. Primary Outcome: Headache Days as Self-reported by Participants
Description: At the seven day follow-up, participants will be asked by phone how many days they experienced headaches since being discharged.
Time Frame: 7 days after discharge from emergency department
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Control | Experimental
Number analyzed (Participants) | 101 | 106
days | 3.0 [2.5 to 3.5] | 3.3 [2.8 to 3.9]

2. Secondary Outcome: Number of Participants With Sustained Headache Freedom
Description: Sustained headache freedom is defined as achieving a headache intensity = none within two hours of treatment and maintaining this level, without requiring additional headache medication, for 7 days following discharge from the Emergency Department. Participants will be asked by phone how number of days they experienced headaches during the week after discharge from the emergency department. Reported values are participants who experienced no headaches at all during the 7 days immediately following discharge.
Time Frame: 7 days after discharge from emergency department
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 107 | 110
Participants | 10 | 6

3. Secondary Outcome: Medication Preference as Assessed by Self-report
Description: Participants will be asked, by phone, if they would want the same medication during a subsequent visit to the emergency department. Reported values indicate participants who responded "yes".
Time Frame: 7 days after discharge from emergency department
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 101 | 106
Participants | 76 | 75

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Control | Experimental
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/111
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/111
Other Adverse Events (participants affected / at risk) | 3/109 | 16/111
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=109) | Experimental (N=111)
Akathisia (Nervous system disorders) | 2 (2) | 7 (7)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT02847494/Prot_SAP_000.pdf